CLINICAL TRIAL: NCT05081609
Title: IL Believe: A Phase 1/2, Open-label, Dose Escalation and Dose Expansion Study to Investigate the Safety and Tolerability of TransCon IL-2 β/γ Alone or in Combination With Pembrolizumab, TransCon TLR7/8 Agonist, or Other Anticancer Therapies, in Adult Participants With Locally Advanced or Metastatic Solid Tumor Malignancies
Brief Title: A Study to Investigate Safety and Tolerability of TransCon IL-2 β/γ Alone or in Combination With Pembrolizumab and/or TransCon TLR7/8 Agonist or Other Anticancer Therapies in Adult Participants With Locally Advanced or Metastatic Solid Tumor Malignancies
Acronym: IL Believe
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ascendis Pharma Oncology Division A/S (Industry)
Responsible Party: Sponsor
Organization: Ascendis Pharma A/S (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ASND0029
Record Dates: First submitted 2021-10-05; First posted 2021-10-18 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumor; Locally Advanced Solid Tumor; Metastatic Solid Tumor; Platinum-resistant Ovarian Cancer; Post Anti-PD-1 Melanoma; 2L+ Cervical Cancer; Neoadjuvant Melanoma; Neoadjuvant Non-Small Cell Lung Cancer; Post Anti-PD-(L)1 Non-Small Cell Lung Cancer; Post Anti-PD-(L)1 Small Cell Lung Cancer; Third Line or Later (3L+) HER2+ Breast Cancer; Second or Third Line (2L/3L) Cervical Cancer; Third-line or Later (3L+) Platinum-resistant Ovarian Cancer (PROC)
MeSH Terms: conditions — Neoplasm Metastasis; Uterine Cervical Neoplasms | interventions — pembrolizumab; Surgical Procedures, Operative; Trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part 1 Monotherapy Dose Escalation: TransCon IL-2 β/γ (Experimental): TransCon IL-2 β/γ in escalating doses to evaluate safety/tolerability and to determine the MTD and RP2D
  Interventions: Drug: TransCon IL-2 β/γ
- Part 2 Combination Dose Escalation: TransCon IL-2 β/γ with Pembrolizumab (Experimental): TransCon IL-2 β/γ with Pembrolizumab in escalating doses to evaluate safety/tolerability and determine the MTD and RP2D
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Pembrolizumab
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with SOC Chemo (Experimental): TransCon IL-2 β/γ using the RP2D with SOC Chemotherapy to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Chemotherapy drug
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with TransCon TLR7/8 Agonist (Experimental): TransCon IL-2 β/γ with TransCon TLR7/8 Agonist using the RP2D to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Drug: TransCon TLR7/8 Agonist
- Part 3 Monotherapy Dose Expansion: TransCon IL-2 β/γ followed by surgery (Experimental): (Optional Arm): TransCon IL-2 β/γ using the RP2D followed by surgery to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Procedure: Surgery
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with Pembrolizumab followed by surgery (Experimental): TransCon IL-2 β/γ using the RP2D with Pembrolizumab followed by surgery to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Pembrolizumab; Procedure: Surgery
- Part 3 Combination Dose Expansion:TransCon IL-2 β/γ with TransCon TLR7/8 Agonist followed by surgery (Experimental): TransCon IL-2 β/γ with TransCon TLR7/8 Agonist using the RP2D followed by surgery to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Drug: TransCon TLR7/8 Agonist; Procedure: Surgery
- Part 3 Combination Dose Expansion:TransCon IL-2 β/γ + Pembrolizumab + SOC Chemo followed by surgery (Experimental): TransCon IL-2 β/γ using the RP2D with Pembrolizumab and SOC Chemotherapy followed by surgery to evaluate safety/tolerability and anti-tumor activity of the combination
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Pembrolizumab; Drug: Chemotherapy drug; Procedure: Surgery
- Part 3 Combination Dose Expansion (Experimental): TransCon IL-2 β/γ + Pembrolizumab TransCon IL-2 β/γ using the RP2D with Pembrolizumab
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Pembrolizumab
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ monotherapy (Experimental): TransCon IL-2 β/γ monotherapy
  Interventions: Drug: TransCon IL-2 β/γ
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ + trastuzumab (Experimental): TransCon IL-2 β/γ + trastuzumab
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Trastuzumab
- Part 3 Combination Dose Expansion: TransCon IL-2 β/γ + trastuzumab emtansine (T-DM1) (Experimental): TransCon IL-2 β/γ + trastuzumab emtansine (T-DM1)
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Trastuzumab emtansine (T-DM1)
- Part 4 Combination Dose Optimization (Experimental): TransCon IL-2 β/γ + Pembrolizumab TransCon IL-2 β/γ using the RP2D in titrating doses and/or different dose frequencies with Pembrolizumab
  Interventions: Drug: TransCon IL-2 β/γ; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TransCon IL-2 β/γ — TransCon IL-2 β/γ will be administered as an intravenous (IV) infusion
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous (IV) infusion
  Arms: Part 2 Combination Dose Escalation: TransCon IL-2 β/γ with Pembrolizumab; Part 3 Combination Dose Expansion; Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with Pembrolizumab followed by surgery; Part 3 Combination Dose Expansion:TransCon IL-2 β/γ + Pembrolizumab + SOC Chemo followed by surgery; Part 4 Combination Dose Optimization
Drug: Chemotherapy drug — SOC chemotherapy will be administered as an intravenous (IV) infusion
  Arms: Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with SOC Chemo; Part 3 Combination Dose Expansion:TransCon IL-2 β/γ + Pembrolizumab + SOC Chemo followed by surgery
Drug: TransCon TLR7/8 Agonist — TransCon TLR7/8 Agonist will be administered as an IT (Intratumoral) injection
  Arms: Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with TransCon TLR7/8 Agonist; Part 3 Combination Dose Expansion:TransCon IL-2 β/γ with TransCon TLR7/8 Agonist followed by surgery
Procedure: Surgery — Surgery will take place 4-6 weeks after last dose of study treatment.
  Arms: Part 3 Combination Dose Expansion: TransCon IL-2 β/γ with Pembrolizumab followed by surgery; Part 3 Combination Dose Expansion:TransCon IL-2 β/γ + Pembrolizumab + SOC Chemo followed by surgery; Part 3 Combination Dose Expansion:TransCon IL-2 β/γ with TransCon TLR7/8 Agonist followed by surgery; Part 3 Monotherapy Dose Expansion: TransCon IL-2 β/γ followed by surgery
Drug: Trastuzumab — Trastuzumab will be administered as an intravenous (IV) infusion
  Arms: Part 3 Combination Dose Expansion: TransCon IL-2 β/γ + trastuzumab
Drug: Trastuzumab emtansine (T-DM1) — Trastuzumab emtansine (T-DM1) will be administered as an intravenous (IV) infusion
  Arms: Part 3 Combination Dose Expansion: TransCon IL-2 β/γ + trastuzumab emtansine (T-DM1)

SUMMARY:
TransCon IL-2 β/γ is an investigational drug being developed for treatment of locally advanced or metastatic solid tumors. This is a first-in-human, open-label, Phase 1/2, dose escalation and dose expansion study of TransCon IL-2 β/γ as monotherapy or in combination therapy in adult participants with advanced or metastatic solid tumors. Given the unique PK profile enabled by the TransCon technology, TransCon IL-2 β/γ presents the opportunity to enhance the therapeutic index of current IL-2 therapy.

DETAILED DESCRIPTION:
IL-2 is a key cytokine that directs the immune system through pleiotropic effects mediated by promoting expansion of both cytotoxic effector cells and Tregs. TransCon IL-2 β/γ is designed as a long-acting delivery prodrug of IL-2 β/γ, a potent cytokine signaling molecule, with the potential to improve the safety and efficacy of IL-2.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years of age, or country defined local legal age
* Demonstrated adequate organ function at screening
* Life expectancy >12 weeks as determined by the Investigator
* Female and male participants of childbearing potential who are sexually active must agree to use highly effective methods of contraception
* Participants must have histologically confirmed locally advanced, recurrent, or metastatic solid tumor malignancies that cannot be treated with curative intent (surgery or radiotherapy), with the exception of the neoadjuvant cohorts
* Part 1 and Part 2: Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Part 3 and Part 4: Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Participants who have undergone treatment with anti-PD-1, anti-PD-L1, or anti-cytotoxic T-lymphocyte-associated protein (CTLA-4) antibody must have a washout of at least 4 weeks from the last dose and evidence of disease progression per investigator assessment before Cycle 1 Day 1 (C1D1) with the exception of the neoadjuvant cohorts
* Participants who have previously received an immunotherapy prior to C1D1 must have any immune-related toxicities resolved to ≤Grade 1 or baseline (prior to the immunotherapy) to be eligible, with the exception of participants on well controlled physiologic endocrine replacement
* Part 3: Neoadjuvant cohorts: participants must have completely resectable disease

Key Exclusion Criteria:

* Symptomatic central nervous system metastases and/or carcinomatous meningitis
* Active autoimmune diseases, regardless of need for immunosuppressive treatment, with the exception of participants well controlled on physiologic endocrine replacement
* Any uncontrolled bacterial, fungal, viral, or other infection
* Significant cardiac disease
* A marked clinically significant baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >480 ms) [CTCAE Grade 1]) using Fridericia's QT correction formula
* Positive for human immunodeficiency virus (HIV) or has known active hepatitis B or C infection
* Known hypersensitivity to any study treatment(s) used in the specific study part/cohort
* Participants who have been previously treated with IL-2 or IL-2 variants (all participants)
* Systemic immunosuppressive treatment with the exception for patients on corticosteroid taper (for example, for chronic obstructive pulmonary disease exacerbation).
* Vaccination with live, attenuated vaccines within 4 weeks of C1D1
* Treatment with any other anti-cancer systemic treatment (approved or investigational) or radiation therapy within 4 weeks of C1D1
* Part 3: Other active malignancies within the last 2 years
* Women who are breastfeeding or have a positive serum pregnancy test during screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Through study completion, expected average of 2 years
  Treatment emergent and treatment related adverse events (assessed by NCI CTCAE v5.0), serious adverse events (SAEs), adverse events leading to treatment discontinuation, deaths.
Maximum Tolerated Dose (MTD) | Each cycle is 21 days
  Determine the maximum tolerated dose by assessing the Incidence of Dose Limiting Toxicities (DLTs), treatment emergent and treatment related adverse events (assessed by NCI CTCAE v5.0), serious adverse events (SAEs), adverse events leading to treatment discontinuation and deaths.
Recommended Phase 2 Dose (RP2D) | 12 months
  To determine a recommended phase 2 dose of TransCon IL-2 β/γ and combination regimen for further development by evaluating number of patients with treatment-related adverse events as assessed by CTCAE.

SECONDARY OUTCOMES:
Overall Response Rate | Average of 2 years
  Response assessed by RECIST v1.1
Pathologic Complete Response | 15 weeks
  Evaluate the pathologic Complete Response (pCR) for anti-tumor activity of TransCon IL-2 β/γ alone or in combination with pembrolizumab, or TransCon TLR7/8 Agonist, or in combination with pembrolizumab and SOC chemotherapy in the Neoadjuvant Cohorts
Major Pathologic Response | 15 weeks
  Evaluate the Major Pathologic Response (MPR) for anti-tumor activity of TransCon IL-2 β/γ alone or in combination with pembrolizumab, or TransCon TLR7/8 Agonist, or in combination with pembrolizumab and SOC chemotherapy in the Neoadjuvant Cohorts
Duration of Response | Average of 2 years
  Time from first documentation of objective tumor response (CR or PR that is subsequently confirmed) to first documentation of disease progression or death due to any cause, whichever occurs first
Time to Response | Expected up to 1 year from first dose
  Time from date of first dose of study treatment to first occurrence of response (CR or PR)
Progression Free Survival (PFS) | Average of 2 years
  Time from date of first dose of study treatment to first documentation of disease progression or death due to any cause
Event free survival (EFS) by RECIST 1.1 | 2 years
  Time from the date of the first dose of study treatment to the occurrence of any of the following: progression of disease that precludes surgery, disease recurrence after surgery, or death from any cause.
Overall Survival (OS) | Average of 2 years
  Time from date of first dose of study treatment to date of death due to any cause
PK Characterization (Cmax) | Average of 2 years
  Maximum observed plasma concentration of TransCon IL-2 β/γ and Free IL-2 β/γ after IV administration of TransCon IL-2 β/γ alone or in combination with other therapies
PK Characterization (Tmax) | Average of 2 years
  Time to reach maximum plasma concentration of TransCon IL-2 β/γ and Free IL-2 β/γ after IV administration of TransCon IL-2 β/γ alone or in combination other therapies
PK Characterization (AUClast) | Average of 2 years
  Area under the plasma concentration curve from time zero to last sampling time at which the concentration is at or above the lower limit of quantification for TransCon IL-2 β/γ and Free IL-2 β/γ after IV administration of TransCon IL-2 β/γ alone or in combination with other therapies
PK Characterization (AUC0-t) | Average of 2 years
  Area under the plasma concentration curve from time zero to time t for TransCon IL-2 β/γ and Free IL-2 β/γ after IV administration of TransCon IL-2 β/γ alone or in combination with other therapies
PK Characterization (t1/2) | Average of 2 years
  Apparent terminal half-life of TransCon IL-2 β/γ and Free IL-2 β/γ after IV administration of TransCon IL-2 β/γ alone or in combination with other therapies

CONTACTS AND LOCATIONS:
Overall Officials: Davis Torrejon-Castro, Study Director — Medical Monitor
Locations (51):
- United States (13):
  - Ascendis Pharma Investigational Site, Los Angeles, California
  - Ascendis Pharma Investigational Site, Springfield, Illinois
  - Ascendis Pharma Investigational Site, Louisville, Kentucky
  - Ascendis Pharma Investigational Site, Boston, Massachusetts
  - Ascendis Pharma Investigational Site, Morristown, New Jersey
  - Ascendis Pharma Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Huntersville, North Carolina
  - Ascendis Pharma Investigational Site, Canton, Ohio
  - Ascendis Pharma Investigational Site, Cincinnati, Ohio
  - Ascendis Pharma Investigational Site, Oklahoma City, Oklahoma
  - Ascendis Pharma Investigational Site, Pittsburgh, Pennsylvania
  - Ascendis Pharma Investigational Site, Nashville, Tennessee
  - Ascendis Pharma Investigational Site, Richmond, Virginia
- Australia (6):
  - Ascendis Pharma Investigational Site, Adelaide
  - Ascendis Pharma Investigational Site, Brisbane
  - Ascendis Pharma Investigational Site, Frankston
  - Ascendis Pharma Investigational Site, Southport
  - Ascendis Pharma Investigational Site, Toorak Gardens
  - Ascendis Pharma Investigational Site, Waratah
- Ascendis Pharma Investigational Site, Wilrijk, Belgium
- Canada (2):
  - Ascendis Pharma Investigational Site, Montreal
  - Ascendis Pharma Investigational Site, Toronto
- Italy (12):
  - Ascendis Pharma Investigational Site, Cuneo
  - Ascendis Pharma Investigational Site, Florence
  - Ascendis Pharma Investigational Site, Grosseto
  - Ascendis Pharma Investigational Site, Lido di Camaiore
  - Ascendis Pharma Investigational Site, Livorno
  - Ascendis Pharma Investigational Site, Meldola
  - Ascendis Pharma Investigational Site, Milan
  - Ascendis Pharma Investigational Site, Modena
  - Ascendis Pharma Investigational Site, Roma
  - Ascendis Pharma Investigational Site, Torino
  - Ascendis Pharma Investigational Site, Turin
  - Ascendis Pharma Investigational Site, Verona
- Poland (3):
  - Ascendis Pharma Investigational Site, Krakow
  - Ascendis Pharma Investigational Site, Poznan
  - Ascendis Pharma Investigational Site, Warsaw
- Ascendis Pharma Investigational Site, Singapore, Singapore
- South Korea (3):
  - Ascendis Pharma Investigational Site, Seoul, Songpa-gu
  - Ascendis Pharma Investigational Site, Seongnam-si
  - Ascendis Pharma Investigational Site, Seoul
- Spain (9):
  - Ascendis Pharma Investigational Site, Barcelona
  - Ascendis Pharma Investigational Site, L'Hospitalet de Llobregat
  - Ascendis Pharma Investigational Site, Madrid
  - Ascendis Pharma Investigational Site, Málaga
  - Ascendis Pharma Investigational Site, Murcia
  - Ascendis Pharma Investigational Site, Oviedo
  - Ascendis Pharma Investigational Site, Pamplona
  - Ascendis Pharma Investigational Site, Seville
  - Ascendis Pharma Investigational Site, Valencia
- Ascendis Pharma Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rosen DB, Kvarnhammar AM, Laufer B, Knappe T, Karlsson JJ, Hong E, Lee YC, Thakar D, Zuniga LA, Bang K, Sabharwal SS, Uppal K, Olling JD, Kjaergaard K, Kurpiers T, Schnabel M, Reich D, Glock P, Zettler J, Krusch M, Bernhard A, Heinig S, Konjik V, Wegge T, Hehn Y, Killian S, Viet L, Runz J, Faltinger F, Tabrizi M, Abel KL, Breinholt VM, Singel SM, Sprogoe K, Punnonen J. TransCon IL-2 beta/gamma: a novel long-acting prodrug with sustained release of an IL-2Rbeta/gamma-selective IL-2 variant with improved pharmacokinetics and potent activation of cytotoxic immune cells for the treatment of cancer. J Immunother Cancer. 2022 Jul;10(7):e004991. doi: 10.1136/jitc-2022-004991. PMID 35817480